CLINICAL TRIAL: NCT04339374
Title: Diagnosis and Risk Assessment of Locally Advanced Rectal Cancer Using Co-registered Ultrasound and Photoacoustic Imaging
Brief Title: Ultrasound and Photoacoustic Imaging for Enhanced Differential Diagnosis of Rectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201707066; 1R01EB034398 (NIH)
Record Dates: First submitted 2020-03-30; First posted 2020-04-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Rectal Cancer; Colorectal Cancer
Keywords: Rectal cancer; Nonoperative management; Watch and wait; Complete clinical response
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- In vivo imaging (Other): * Patients with distal rectal lesions (benign or malignant tumors within 15cm of the anal verge) will be enrolled for the in vivo imaging portion of the study
  * Participation will include an intraoperative, in vivo evaluation of the tumor with a novel endorectal photoacoustic ultrasound probe. Following the induction of anesthesia, patients will undergo a 20-minute endorectal imaging evaluation performed by their colorectal surgeon. After imaging, the patient will then undergo standard-of-care surgical resection of the rectum. The resection specimen may then be imaged ex vivo as deemed necessary.
  * For this portion of the study, enrollment will be limited to a total of 86 participants
  Interventions: Device: Photoacoustic imaging, photoacoustic microscopy; Device: Endorectal photoacoustic imaging probe
- Reader Team (Experimental): 3 surgeons and 1 radiologist will be initially trained to grade lesions using the PAM/US image from the first set of 30 patients (Group 1). They will then use the PAM/US data to grade lesions obtained from the second set of 56 patients after initial training (Group 2).
  Interventions: Device: Photoacoustic imaging, photoacoustic microscopy; Device: Endorectal photoacoustic imaging probe; Other: Reader Performance

INTERVENTIONS:
Device: Photoacoustic imaging, photoacoustic microscopy — -Emerging technique in which a short-pulsed laser beam penetrates diffusely into a tissue sample, causing the release of acoustic waves due to a transient temperature rise -The transient acoustic waves, or photoacoustic waves, are then measured around the sample by US transducers -The resolution of the devices can be altered by changing the wavelengths of laser light and spectrum analysis of the receiver. In this manner, human colorectal pathology will be examined under multiple types of photoacoustic ranges (broadly termed photoacoustic microscopy and photoacoustic imaging). The study has two phases. In the second phase, the investigators will provide assessments of treated rectum based on clinical information and photoacoustic information after initial training.
  Other Names: PAI; PAM
Device: Endorectal photoacoustic imaging probe — -An endorectal imaging device using coregistered photoacoustic and ultrasound imaging has been constructed. This probe is used to perform in vivo imaging among patients with rectal pathology intraoperatively.
  Other Names: PAI; Coregistered photoacoustic ultrasound imaging; PAM
Other: Reader Performance — After initial training using Group 1 data, readers will classify lesions as non-clinical complete responders (non-cCR) or clinical complete responders (cCR) based on standard-of-care (SOC) information. Following PAM/US imaging, readers will reassess lesion status using PAM/US data. PAM/US model outputs will be generated for each patient and compared with reader assessments. For patients undergoing surgery, tumor regression scores from surgical specimens will be compared with reader assessments and model outputs. For patients under nonoperative surveillance, clinical response at 2-year follow-up will be compared with model outputs. The study will evaluate whether PAM/US assistance improves residual tumor detection in Group 2 patients. As the model is under development, it will be iteratively retrained and tested as new data become available.
  Arms: Reader Team

SUMMARY:
The purpose of this study is to demonstrate the functionality of a novel endorectal photoacoustic ultrasound imaging modality in humans with rectal cancer. The study involves testing a previously developed endorectal device to determine its ability to accurately assess rectal tumor response to preoperative treatment. Investigators hypothesize that a co-registered photoacoustic ultrasound endorectal device can significantly reduce unnecessary surgeries in rectal cancer patients with complete clinical response while maintaining high sensitivity in identifying those with residual cancer.

DETAILED DESCRIPTION:
The investigators hypothesize that a co-registered photoacoustic ultrasound endorectal device can significantly reduce unnecessary surgeries in rectal cancer patients with complete clinical response while maintaining high sensitivity in identifying those with residual cancer. The proposed new imaging technique combined with deep-learning algorithms will provide a real-time imaging tool to assist surgeons in predicting the neoadjuvant treatment response of rectal cancer patients. Such a tool will offer sensitive vascular and %sO2 contrast for identifying complete responses, thereby assisting surgeons in significantly improving sensitivity and specificity in surgery recommendations. The study will 1) rigorously validate the technique in a group of locally advanced rectal cancer (LARC) patients who will undergo surgical resection or "wait and watch" surveillance of their rectum based on the standard of care (SOC), and 2) explore the technique's potential in assessing a sub-group of LARC patients through the course of neoadjuvant treatment and in post-treatment surveillance. Successful completion of the project will result in a new imaging tool that can significantly improve the SOC by reducing unnecessary surgery without compromising cancer-related outcomes and thereby lowering morbidity and health care cost.

In this trial, the investigators will recruit patients with rectal cancer who have completed neoadjuvant therapy and will undergo surgery or nonoperative management. Approximately 86 patients will be recruited. The first group of 30 patients (group #1) will be used to train/validate identification algorithm. The second group of 56 patients (group #2) will be used as the testing cohort to train the reader team comprised of 3 surgeons and 1 radiologist. Eligible patients will include those with rectal cancer who received neoadjuvant therapy and were deemed to either have incomplete or indeterminant or clinical response based on standard endoscopy and axial imaging with magnetic resonance. PAM/US will be performed before their surgery or at the time of patients' follow up imaging.

In the investigation of group #2 patients, the study surgeon will review each patient's record and decide on surgery (clinical non-responders, non-cCR) for two types of patients of 1) those deemed non-cCR based on SOC at the treatment completion; 2) those deemed cCR at the treatment completion and are under "watch and wait" surveillance .

After initial training using group #1 data, the study surgeon will grade the tumor bed based on MRI and other clinical information as non-cCR or cCR at the time of SOC imaging after treatment completion. PAM/US imaging will be performed at the same time as the patients' SOC imaging. The study surgeon will grade the tumor bed as either PAM/US non-cCR or PAM/US cCR after PAM/US imaging.

For patients with surgery, the pathological outcomes of the patients will be assessed based on the Modified Ryan Scheme for Tumor Regression Score. Score 0, No viable cancer cells (pCR); Score 1, Single cells or rare small groups of cancer cells (near pCR); Score 2, Residual cancer with evident tumor regression, but more than single cells or rare small groups of cancer cells; Score 3, Extensive residual cancer with no evident tumor regression. Scores 2 and 3 are considered as non-pCRs. For patients without surgery, cCR without of any concerns of recurrence at the end of 2 year follow-up window will be considered as responder. The radiologist reader will also independently grade each case based on MRI.

The sensitivity and specificity as well as the area under the receiver operation characteristic curve (AUC) of the reader team based on the SOC will be evaluated. The sensitivity and specificity and AUC of the reader team based on PAM/US data will be evaluated. If the PAM/US methodology is validated from this prospective study, surgeries could be reduced in this group of patients who are pCRs or near pCRs and whose PAM/US imaging scores provided by reader team classify them as responders. PAM/US-model outputs will be computed for each patient and compared with reader's assessment . The investigators will also correlate MRI/DWI findings with PAM/US and document agreement/discordance with explanations.

As an exploratory part of this trial, a subset of eligible patients of group #2 of will be selected to undergo three serial imaging studies: at pre-treatment, halfway through treatment (after completion of one week of radiation followed by 2 months of chemotherapy), and at treatment conclusion (after one week of radiation followed by 4 months of chemotherapy). At the treatment conclusion, those deemed to have residual tumor by standard clinical methods (~65%) will proceed to surgery. For the remaining 35% of patients, with no evidence of active disease, surveillance will be initiated. For these patients, serial imaging examinations will be performed every six months (coordinated with standard examinations). Patients deemed to have a recurrence will undergo surgery.

Once every enrolled patient in this subgroup has completed either surgery or two years of surveillance, the participants will be divided into two groups: Group A (those who underwent surgery) and Group B (those treated solely with nonoperative surveillance). As the primary outcome, Group A will demonstrate the accuracy of photoacoustic imaging. As a secondary outcome, Group A will reveal how the tumor vasculature and %sO2 changes over time, which may provide new insight into how complete response patients respond differently from non-pCR patients and how PAM/US can capture these earlier changes. The investigators will follow up on their SOC results in the clinical system and correlate their PAM/US results during the 2-year surveillance with their five-year disease-free survival.

To identify each patient as a complete or non-complete responder, the investigators will analyze photoacoustic images of all group #2 56 patients serially with the reader team assisted by PAM/US models developed earlier in the trial. These quantitative measures, as well as any qualitative local vasculature and %sO2 changes and US morphological changes, will be recorded at each time point. Standard MRI and endoscopic images will be independently collected and analyzed. Since the novel PAM/US model is in the development stage, the investigators may need to continuously re-train the model with more data collected and test the model from new cases to improve the model performance.

As a final part of this trial, the investigators will explore patterns of post-treatment vascular and %sO2 changes during preoperative treatment and serial surveillance. Tumor angiogenesis in colorectal cancer has been well studied using microvessel density (MVD) as a surrogate marker. While high levels of MVD and vascular endothelial growth factor (VEGF) significantly predict poor survival, little is known about the dynamics of vascular and %sO2 changes and the mechanisms of neovascularization after chemoradiation.

The investigators have observed tumor beds revert from oncologically-disrupted microvascular patterns to highly regular architecture typical of the normal rectum where pCR has occurred, though this mechanism is not well-understood. In contrast, heterogeneous and often microvascular-deficient regions have been found consistently in tumor beds with residual cancer at treatment completion. This novel imaging device could serve as a new platform for investigating the dynamics of vascular and %sO2 changes during and after therapy and for assessing potential rectal cancer recurrence early on. In addition to PAM/US imaging studies, the surgeon will perform biopsies at the central region and edges of the tumor bed before treatment, at treatment completion (if no surgery), and at the point of tumor reoccurrence. For patients with surgery, surgical samples will be used. Specifically, MVD and VEGF expression will be assessed by immunohistochemical staining, and both will be quantitatively correlated with PAM/US findings at the center of the tumor bed and at the tumor edges. The results will help the investigators understand how vasculature changes during treatment and at recurrence are correlated with imaging findings.

ELIGIBILITY:
Inclusion Criteria Patients:

* Patients with any stage of rectal cancer undergoing surgical resection.
* Age >18 years
* Able to provide informed consent

Additional Inclusion Criterion for in vivo imaging (patients):

* Lesion located within 15cm of the anal verge

Exclusion Criteria Patients:

* Inability to provide consent
* Collection of intraoperative specimen for frozen section analysis will disqualify patients from participation

Eligibility Criteria Readers:

* Colorectal surgeons or radiologists who treat or interpret imaging regularly for patients with rectal cancer.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients that readers are able to diagnose with rectal cancer | Approximately 15 minutes
  The primary endpoint is to see if the readers trained to use the co-registered PAM/US data are able to diagnose rectal cancers with better sensitivity & specificity using surgery pathology results as the ground truth.
  SOC sensitivity and specificity will be computed based on readers' cCR vs. non-cCR. The sensitivity and specificity with additional PAM/US data will be computed based on readers' revised cCR vs. non-cCR. PAM/US model sensitivity and specificity will also be computed using surgery pathology results.
Number of patients without surgery who cleared as cCR after 2-years of follow-up | 2-years of follow-up
  The secondary primary endpoint is the sensitivity and specificity of readers' cCR vs. non-cCR assessments using SOC and sensitivity and specificity of PAM/US models cCR vs. non-cCR reassessments PAM/US data. The "ground truth " of this cohort will be no cancer recurrence based on clinical data.

SECONDARY OUTCOMES:
Area under the receiver operating curve (ROC) | Approximately 15 minutes
  The secondary outcome is the accuracy of co-registered PAM/US in assisting surgeons on risk management and surgery recommendation by measuring the area under the receiver operating curve (AUC) in a cohort of patients with the designed statistical power given in the power analysis.
Characterize in vivo tissue samples with photoacoustic imaging | Approximately 15 minutes
  This outcome will be measured qualitatively by comparing histologic (ex vivo) findings to the experimental imaging. The critical features to be analyzed in each image are the cross-sectional structure of normal colorectal tissues in comparison to the loss of a layered structure and its corresponding evenly distributed vascular pattern in the setting of neoplasia.
Performance characteristics of the novel endorectal ultrasound probe as measured by number of adverse events | Approximately 15 minutes
Performance characteristics of the novel endorectal ultrasound probe as measured by evidence of tissue damage from the imaging laser | Approximately 15 minutes
Performance characteristics of the novel endorectal ultrasound probe as measured by time required to complete study | Approximately 15 minutes
Performance characteristics of the novel endorectal ultrasound probe as measured by variability in image production | Approximately 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: William Chapman, Jr., M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
* Data available for sharing - Code and de-identified patient data related to this project will be made available upon request to other academic entities following the publication of project-related results.
  * Data to be shared - Individual participant data, along with code related to the novel neural network developed, that underlie the results reported herein. Data will not be shared until deidentified.
  * With whom will data be shared - academic entities approved by the primary research team
Supporting Information: Study Protocol
Time Frame: Data will be made available to approved persons between 12 and 36 months after publication of these results
Access Criteria: * Purpose of accessing data - any purpose allowed.
  * Mechanism for sharing data - data to be shared via institutional file sharing service once appropriate parties have been approved by the research team.

REFERENCES:
- [Derived] Leng X, Uddin KMS, Chapman W Jr, Luo H, Kou S, Amidi E, Yang G, Chatterjee D, Shetty A, Hunt S, Mutch M, Zhu Q. Assessing Rectal Cancer Treatment Response Using Coregistered Endorectal Photoacoustic and US Imaging Paired with Deep Learning. Radiology. 2021 May;299(2):349-358. doi: 10.1148/radiol.2021202208. Epub 2021 Mar 23. PMID 33754826
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu